CLINICAL TRIAL: NCT04798469
Title: Androgen Replacement to Improve Patient-Important Outcomes in Men With Opioid-Induced Hypogonadism
Brief Title: Pain Alleviation With Testosterone in Opioid-Induced Hypogonadism
Acronym: PATH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shehzad Basaria, M.D., Professor of Medicine, Harvard Medical School; Associate Director, Section on Men's Health, Aging & Metabolism, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P000331
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use; Pain; Hypogonadism, Male
Keywords: Pain; Opioid Analgesics; Testosterone
MeSH Terms: conditions — Pain; Eunuchism | interventions — testosterone undecanoate; Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Experimental): Intramuscular injections of testosterone undecanoate 750 mg.
  Interventions: Drug: Testosterone Undecanoate 250 MG/ML
- Placebo (Placebo Comparator): Intramuscular injections of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone Undecanoate 250 MG/ML — Intramuscular administration at a dose of 750 mg at baseline, weeks 4, and week 14.
  Other Names: Testosterone
  Arms: Testosterone
Drug: Placebo — Intramuscular administration of placebo at baseline, weeks 4, and week 14.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The aim of this trial is to evaluate whether testosterone replacement results in greater improvement in pain perception, pain tolerance, sexual function, fatigue, and quality of life when compared with placebo in men with chronic spinal pain treated with opioids who have opioid-induced hypogonadism (low testosterone).

DETAILED DESCRIPTION:
This single-center, randomized, double-blind, placebo-controlled, parallel-group trial will evaluate pain and quality of life outcomes associated with 6 months of treatment with testosterone or placebo in men aged 18 years or older with chronic non-cancer spinal pain who are taking opioid analgesics for at least 6 months and have opioid-induced hypogonadism.

ELIGIBILITY:
Inclusion Criteria:

* Men, age 18 years and older.
* Chronic non-cancer spinal pain.
* Use of opioid analgesics for at least 6 months.
* Serum total testosterone (measured by mass spectrometry) <348 ng/dL and/or free testosterone <70 pg/mL.
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* History of prostate cancer or breast cancer.
* Known history of organic hypogonadism (e.g., due to hypothalamic, pituitary or testicular disease).
* Use of testosterone within the past 6 months.
* Baseline hematocrit >48%.
* Prostate-specific antigen (PSA) level >4 ng/mL in Caucasians or >3 ng/mL in African-Americans.
* Presence of prostate nodule or induration on digital rectal examination.
* Uncontrolled congestive heart failure.
* Myocardial infarction, acute coronary syndrome, revascularization surgery or stroke within 3 months.
* Serum creatinine >2.5 mg/dL.
* Alanine aminotransferase (ALT) level 3 times above the upper limit of normal.
* Diagnosis of bipolar disorder or schizophrenia.
* Presence of metallic implants (pacemakers, aneurysm clips, etc.) that preclude the patient from undergoing functional magnetic resonance imaging (MRI). In subjects who are otherwise eligible and either do not qualify for MRI or are reluctant to undergo imaging, the investigators may consider enrolling such participants on a case-by-case basis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in scores in the Pain Interference Subscale of the Brief Pain Inventory (BPI) questionnaire | Baseline, 3 months, and 6 months
  The Pain Interference Subscale of the BPI is specifically relevant to patients with chronic back pain who are using opioids and correlates strongly with the patient's quality of life.

SECONDARY OUTCOMES:
Changes in response to quantitative sensory testing of pain under pressure stimulus | Baseline, 3 months, and 6 months
  Responses to pressure stimulation (pressure pain threshold) will be evaluated using a digital pressure algometer.
Changes in response to quantitative sensory testing of pain under deep pressure stimulus | Baseline, 3 months, and 6 months
  Response to deep pressure pain will be ascertained using cuff pressure algometry.
Changes in response to quantitative sensory testing of pain under a mechanical stimulus | Baseline, 3 months, and 6 months
  Responses to mechanical pain will be assessed using repetitive stimuli (temporal summation or "windup") with a set of punctate mechanical probes.
Changes in response to quantitative sensory testing of pain under heat stimulus | Baseline, 3 months, and 6 months
  Responses to heat pain will be assessed using a contact thermode that will deliver thermal stimulation to the skin.
Changes in response to quantitative sensory testing of pain under cold stimulus | Baseline, 3 months, and 6 months
  Responses to cold pain will be assessed using a cold pressor task, which involves immersion of the dominant hand in a circulating water bath at a temperature of 4°C.
Changes in default mode network connectivity | Baseline and 6 months
  Patients with chronic pain show increased default mode network (DMN) connectivity to the anterior/mid-insula, a brain region that integrates multiple dimensions of pain, while reduced DMN connectivity to the insula has been significantly associated with pain reduction. In this trial, we plan to determine the influence of testosterone replacement on DMN connectivity by performing functional magnetic resonance imaging (MRI) before and after testosterone/placebo administration and correlate changes in pain with changes in DMN connectivity.

OTHER OUTCOMES:
Changes in quality of life assessed using the 36-Item Short-Form Survey (SF-36) | Baseline, 3 months, and 6 months
  The SF-36 measures eight QOL domains: physical function, bodily pain, vitality, role limitations due to physical problems, general health perceptions, emotional well-being, social function, and role limitations due to emotional problems. The questionnaire also includes a single item that provides an indication of perceived change in health.
Changes in depressive symptoms assessed with the Patient Health Questionnaire-9 (PHQ-9) | Baseline, 3 months, and 6 months
  The PHQ-9 is a validated health questionnaire that will be administered in this trial to evaluate depression among the participants.
Changes in mood and well-being, assessed using the by Positive and Negative Affect Scale (PANAS) affectivity balance scale | Baseline, 3 months, and 6 months
  The PANAS affectivity balance scale includes 10 questions evaluating positive and negative affect.
Changes in energy, assessed with the Hypogonadism Energy Diary (HED) | Baseline, 3 months, and 6 months
  The HED questionnaire is a self-administered instrument that evaluates energy levels in men with hypogonadism.
Changes in sexual function, assessed with the Sexual Arousal, Interest, and Drive (SAID) questionnaire | Baseline, 3 months, and 6 months
  The SAID questionnaire is a five-item self-administered instrument that evaluates the level of thinking about sex, arousal, and rating the level of interest in sex and sex drive in men with hypogonadism.
Changes in fatigue assessed with the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) questionnaire | Baseline, 3 months, and 6 months
  The FACIT-F questionnaire is a self-reported instrument that evaluates fatigue and its impact on daily activities and function.
Changes in catastrophizing assessed with the Pain Catastrophizing Scale (PCS) questionnaire | Baseline, 3 months, and 6 months
  The PCS is a measure of cognitive and affective responses to pain that consists of 13 items assessing the pain catastrophizing domains of rumination, magnification, and helplessness.
Changes in Patient's Global Impression of Change (PGIC) scores | Baseline and 6 months
  The PGIC is a questionnaire that asks how subjects feel their health status has changed at the end of the study compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Shehzad Basaria, MD, Principal Investigator — Brigham and Women's Hospital; Robert R Edwards, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou R, Turner JA, Devine EB, Hansen RN, Sullivan SD, Blazina I, Dana T, Bougatsos C, Deyo RA. The effectiveness and risks of long-term opioid therapy for chronic pain: a systematic review for a National Institutes of Health Pathways to Prevention Workshop. Ann Intern Med. 2015 Feb 17;162(4):276-86. doi: 10.7326/M14-2559. PMID 25581257
- [Background] Von Korff M, Kolodny A, Deyo RA, Chou R. Long-term opioid therapy reconsidered. Ann Intern Med. 2011 Sep 6;155(5):325-8. doi: 10.7326/0003-4819-155-5-201109060-00011. PMID 21893626
- [Background] Aloisi AM, Ceccarelli I, Fiorenzani P. Gonadectomy affects hormonal and behavioral responses to repetitive nociceptive stimulation in male rats. Ann N Y Acad Sci. 2003 Dec;1007:232-7. doi: 10.1196/annals.1286.022. PMID 14993056
- [Background] Fillingim RB, Edwards RR, Powell T. The relationship of sex and clinical pain to experimental pain responses. Pain. 1999 Dec;83(3):419-425. doi: 10.1016/S0304-3959(99)00128-1. PMID 10568849
- [Background] Basaria S. Male hypogonadism. Lancet. 2014 Apr 5;383(9924):1250-63. doi: 10.1016/S0140-6736(13)61126-5. Epub 2013 Oct 10. PMID 24119423
- [Background] Fillingim RB, Edwards RR. The association of hormone replacement therapy with experimental pain responses in postmenopausal women. Pain. 2001 May;92(1-2):229-34. doi: 10.1016/s0304-3959(01)00256-1. PMID 11323144
- [Background] Daniell HW. Hypogonadism in men consuming sustained-action oral opioids. J Pain. 2002 Oct;3(5):377-84. doi: 10.1054/jpai.2002.126790. PMID 14622741
- [Background] Rajagopal A, Vassilopoulou-Sellin R, Palmer JL, Kaur G, Bruera E. Symptomatic hypogonadism in male survivors of cancer with chronic exposure to opioids. Cancer. 2004 Feb 15;100(4):851-8. doi: 10.1002/cncr.20028. PMID 14770444
- [Background] Basaria S, Travison TG, Alford D, Knapp PE, Teeter K, Cahalan C, Eder R, Lakshman K, Bachman E, Mensing G, Martel MO, Le D, Stroh H, Bhasin S, Wasan AD, Edwards RR. Effects of testosterone replacement in men with opioid-induced androgen deficiency: a randomized controlled trial. Pain. 2015 Feb;156(2):280-288. doi: 10.1097/01.j.pain.0000460308.86819.aa. PMID 25599449
- [Background] Huang G, Travison TG, Edwards RR, Basaria S. Effects of Testosterone Replacement on Pain Catastrophizing and Sleep Quality in Men with Opioid-Induced Androgen Deficiency. Pain Med. 2017 Jun 1;18(6):1070-1076. doi: 10.1093/pm/pnw159. PMID 27550959
- [Background] Kregel J, Meeus M, Malfliet A, Dolphens M, Danneels L, Nijs J, Cagnie B. Structural and functional brain abnormalities in chronic low back pain: A systematic review. Semin Arthritis Rheum. 2015 Oct;45(2):229-37. doi: 10.1016/j.semarthrit.2015.05.002. Epub 2015 May 16. PMID 26092329
- [Background] Meints SM, Mawla I, Napadow V, Kong J, Gerber J, Chan ST, Wasan AD, Kaptchuk TJ, McDonnell C, Carriere J, Rosen B, Gollub RL, Edwards RR. The relationship between catastrophizing and altered pain sensitivity in patients with chronic low-back pain. Pain. 2019 Apr;160(4):833-843. doi: 10.1097/j.pain.0000000000001461. PMID 30531308
- [Background] Katz N, Mazer NA. The impact of opioids on the endocrine system. Clin J Pain. 2009 Feb;25(2):170-5. doi: 10.1097/AJP.0b013e3181850df6. PMID 19333165
- [Background] Edwards RR, Dolman AJ, Michna E, Katz JN, Nedeljkovic SS, Janfaza D, Isaac Z, Martel MO, Jamison RN, Wasan AD. Changes in Pain Sensitivity and Pain Modulation During Oral Opioid Treatment: The Impact of Negative Affect. Pain Med. 2016 Oct;17(10):1882-1891. doi: 10.1093/pm/pnw010. Epub 2016 Mar 1. PMID 26933094
- [Background] Frye CA, Seliga AM. Testosterone increases analgesia, anxiolysis, and cognitive performance of male rats. Cogn Affect Behav Neurosci. 2001 Dec;1(4):371-81. doi: 10.3758/cabn.1.4.371. PMID 12467088
- [Background] Forman LJ, Tingle V, Estilow S, Cater J. The response to analgesia testing is affected by gonadal steroids in the rat. Life Sci. 1989;45(5):447-54. doi: 10.1016/0024-3205(89)90631-0. PMID 2770410
- [Background] Daniell HW, Lentz R, Mazer NA. Open-label pilot study of testosterone patch therapy in men with opioid-induced androgen deficiency. J Pain. 2006 Mar;7(3):200-10. doi: 10.1016/j.jpain.2005.10.009. PMID 16516826
- [Background] Aloisi AM, Ceccarelli I, Carlucci M, Suman A, Sindaco G, Mameli S, Paci V, Ravaioli L, Passavanti G, Bachiocco V, Pari G. Hormone replacement therapy in morphine-induced hypogonadic male chronic pain patients. Reprod Biol Endocrinol. 2011 Feb 18;9:26. doi: 10.1186/1477-7827-9-26. PMID 21332999